CLINICAL TRIAL: NCT00819728
Title: Multicenter Phase II Trial of Weekly Taxotere and Irinotecan (CPT-11) in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Trial of Weekly Taxotere and Irinotecan (CPT-11) in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP56976_US1_203
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Irinotecan

ARMS (1):
- Taxotere/Irinotecan (Experimental)
  Interventions: Drug: Docetaxel; Drug: Irinotecan

INTERVENTIONS:
Drug: Docetaxel — 35mg/m2 IV each week for 4 weeks
  Other Names: Taxotere
Drug: Irinotecan — 50mg/m2 IV each week for 4 weeks

SUMMARY:
The main purpose of the study is to determine the activity of the weekly combination of docetaxel (Taxotere) and irinotecan in terms of response rate in subjects with advanced, previously untreated, non-small cell lung cancer. It is also to determine the activity of this combination in terms of response duration, time to progression, median survival, overall survival, and percent one-year survival, as well as the side-effect and toxicity profile of weekly Taxotere and weekly irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* Microscopically or cytologically confirmed non-small cell lung cancer. Histology may include large cell, squamous cell, undifferentiated, or bronchioalveolar carcinoma, or adenocarcinoma, but no small cell or carcinoid.
* Inoperable stage III B or metastatic stage IV NSCLC
* Measurable (bidimensionally) indicator lesion(s) which have not been irradiated.
* No prior systemic chemotherapy. Prior irradiation for NSCLC is permitted, however, the measurable or evaluable non-measurable disease must be completely outside the radiation portal or there must be radiologic proof of progressive disease. If a patient is receiving palliative radiation, other than the chest, to one site at 30 cGy or less, then the patient is eligible and chemotherapy can proceed immediately after palliative RT.
* ECOG performance status 0 or 1 at screening and on the first day of treatment
* Life expectancy = 12 weeks.
* Patients must be > 4 weeks from prior radiation therapy to the pelvis, spine or long bones, and must be recovered from all side effects.
* Patients must be > 3 weeks from prior major surgery, except for a simple biopsy or placement of a venous access device.

Exclusion Criteria:

* No patient may have the following:
* Neutrophils < 1,500/mm3.
* Platelets < 100,000/mm3.
* Serum creatinine >1.8 mg/dL.
* SGOT > 1.5 times the upper limit of normal for institution.
* Total bilirubin > the upper limit of normal for institution.
* Alkaline phosphatase > 5 times the upper limit of normal for institution.
* Pregnant or lactating females or females of childbearing potential not employing adequate contraception.
* History of other malignancy within the last five years which could affect the diagnosis of NSCLC, except basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Current metastatic CNS disease, if present, must have been treated and clinically stable for at least 3 weeks prior to initial Taxotere treatment. Patients with documented meningeal carcinomatosis are not eligible.
* Grade 2 or greater peripheral neuropathy.
* Psychological, familial, sociological or geographical conditions which do not permit weekly medical follow-up and compliance with the study protocol.
* Patients who are medically unstable, including but not limited to active infection, acute hepatitis, gastrointestinal bleeding, uncontrolled cardiac arrhythmias, uncontrolled angina, uncontrolled hypercalcemia, uncompensated congestive heart failure, uncontrolled diabetes, dementia, seizures, superior vena cava syndrome, and patients whose circumstances do not permit completion of the study or the required follow-up.
* Patients with a history of hypersensitivity reaction to products containing Polysorbate 80 (Tween 80).
* Patients requiring concurrent treatment with corticosteroids unless chronic treatment (> 6 months) at low doses (< 20 mg/day of methylprednisolone or equivalent).
* Patients receiving an investigational drug within 3 weeks of registration.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-06; Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Nagarwala, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis US, Bridgewater, New Jersey, United States